CLINICAL TRIAL: NCT01423591
Title: Infliximab Therapy in Patients With Refractory Polymyalgia Rheumatica: a Double Blind Placebo Controlled Trial
Brief Title: Infliximab Therapy in Patients With Refractory Polymyalgia Rheumatica
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario Marqués de Valdecilla (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Principal Investigator, Dr. Vicente Rodri-guez Valverde, Rheumatology, MD, PhD, Hospital Universitario Marqués de Valdecilla
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04578
Record Dates: First submitted 2011-07-19; First posted 2011-08-26 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Polymyalgia Rheumatica
Keywords: Infliximab; polymyalgia rheumatica; refractory; double blind; placebo controlled; trial
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- infliximab (Experimental)
  Interventions: Drug: infliximab
- inactive powder (Placebo Comparator)
  Interventions: Drug: inactive powder

INTERVENTIONS:
Drug: infliximab — Infliximab 5 mg/kg. i.v. at week 0, 2, 6, 14 y 22.
  Other Names: Remicade, anti-TNF monoclonal Therapy
  Arms: infliximab
Drug: inactive powder — Inactive powder. i.v. at week 0, 2, 6, 14 y 22.
  Other Names: placebo
  Arms: inactive powder

SUMMARY:
Rheumatic Polymyalgia(PMR) is a relatively common chronic inflammatory disorder of unknown origin which predominantly develops in elderly subjects and presents with severe pain and stiffness in the neck, shoulder and pelvic girdles, along with increased acute phase reactants. Systemic manifestations such as fever, anorexia and weight loss are characteristic signatures of PMR.

Corticosteroids (CS) constitute the standard treatment of PMR. Although in most patients the symptoms of the disease disappear after one or two years of treatment, a proportion of patients remain CS-dependent with the subsequent CS toxicity. Open label studies have suggested that tumour necrosis factor (TNF) antagonists lead to sustained improvement and CS sparing effect in patients with refractory PMR.

The investigators conducted a randomised, double-blind, placebo controlled trial with infliximab in CS-dependent patients with PMR. Patients with CS-dependent PMR (defined as requiring ≥ 5 mg/day after at least 2 years of treatment to maintain remission or ≥ 7.5 mg/day after at least 6 months) were randomly assigned to receive Infliximab (5 mg/kg i.v) at 0, 2, 6, 14 and 22 weeks (n = 12) or placebo (n = 11) together with CS that were reduced according to a predefined schedule. The primary outcome was the proportion of responder patients -defined as individuals with both complete clinical and analytical remission without receiving CS for at least three months- at 24 weeks. Secondary outcomes were cumulative CS doses and adverse events proportion.

DETAILED DESCRIPTION:
The duration of the study will be 1 year, and it will be divided in several phases:

A) Initial phase (double-blind trial): Between week 0 and week 24. Placebo or Infliximab at a dose of 3 mg/kg/day at weeks 0, 2 and 6.

After the screening process, patients who meet the inclusion/exclusion criteria of the protocol will be randomized to receive three infusions of placebo or infliximab as previously described.

After the first infusion (week 0), the prednisone dose will be tapered according to the following schedule: Prednisone (or equivalent) should be decreased at a rate of 1.25 mg per week until complete withdrawal of corticosteroids. In case of relapse, the dose of prednisone will be increased up to the previous dose that controlled the symptoms of PMR, and after 4 weeks of stable dose, prednisone will be again tapered but with a slower schedule: 1.25 mg every 2 weeks until complete withdrawal of corticosteroids. In case of a new relapse, the dose of prednisone will be managed according to the physician criteria.

B) Extension phase (open trial): Between week 24 and week 48. Infliximab at a dose of 3 mg/kg/day at weeks 24, 26 and 30.

At 24 weeks, all the patients included into the trial and still on corticosteroid therapy with or without clinical manifestations of PMR, will receive three infusions of infliximab according to the previous described schedule.

After the first infusion (week 24) the dose of prednisone will be decreased according to the same schedule previously described in the initial phase of the trial.

The schedule therapy proposed in the extension phase is going to be for:

* (GROUP A) To evaluate time response to Infliximab in responders concerning active treatment group in phase 1.
* (GROUP B). To incorporate patients placebo- treated to treatment who have showed efficacy (in case of favorable results in the interim analysis)
* (GROUP C). To offer maintenance treatment to patients who have showed complete response during phase 1 and this treatment is associated to a significant corticosteroid tapering dose or maintenance response.
* (GROUP D). Discontinuation of the treatment in patients who have been receiving active treatment during phase 1 and have not showed response in any time.

After the first infusion (week 24), it will be reduced prednisone dose following same regimen described in the clinical phase of the study.

Treatment duration.

•Study will be administrate for 24 + 24 weeks. In the end of the study the patient will continue treatment the most efficacy in the investigator opinion.

Objectives:

Primary objective: Proportion of responders (complete remission without corticosteroids) at 24 weeks.

Secondary objectives:

* Proportion of responders at 48 weeks.
* Time to response
* Number of relapses / recurrences.
* Response duration
* Cumulative dose and side effects of steroids at 24 and 48 weeks.
* Number of patients that should be re-treated with infliximab.
* Side effects of Infliximab in this patient population.
* Serum cytokine analysis

I) CLINICAL ASSESSMENT:

Evaluations will be performed at screening, baseline, every 2 weeks during the first 2 months of treatment and monthly thereafter.

The following data will be recorded at each visit:

* A structured questionnaire on symptoms of PMR.
* Global evaluation of disease activity by the patients and physicians (visual analogue scale, 0-100).
* Global evaluation of pain by the patients (visual analogue scale, 0-100).
* Acute phase reactants: ESR (Westergren) and CRP (nephelometry).
* Complete blood cell count, glucose (glycosylated hemoglobin in case of diabetes), blood urea and creatinine, liver enzymes and albumin.
* Steroid dosage. Cumulative steroid dosage during the study period.
* Presence of relapse
* Side effects, with special emphasis in infections and corticosteroid side effects.

All patients will have a PPD test and chest X-rays performed at screening following the current recommendations for anti-TNF therapy (50-52). Those patients with a positive PPD test (induration ≥ 5 mm) or with chest X-ray images showing lesions consistent with latent tuberculosis infection, will have prophylactic treatment with isoniazid, 300 mg daily during 9 months (in case of isoniazid toxicity: rifamycin, 600 mg/day during four months).

In addition, the patients will be instructed to the possible development of infections and other side effects, and new manifestations of GCA, which should be immediately reported to the attending physician.

II) SERUM CYTOKINE STUDY During the study period and after informed consent, patients will be asked to provide a serum sample (around 200 ml) at 7 different time points (week 0 or pre-treatment, and weeks 2, 6, 24, 26, 30 and 48). The blood will be obtained at the same time that the scheduled venipuncture for routine tests.

The analysis will be done using a Cytometric Bead Array (CBA) methodology. The investigators will use the CBA Flex Set system (Becton Dickinson) that includes the following cytokines: IL-1, IL-6, TGF-beta, TNF-alfa, IL-10, IL-12, IL-2, IL-4, IFN-gamma. Following acquisition of sample data using the FACSCalibur flow cytometer (Becton Dickinson), the sample results are generated in graphical and tabular format using the CBA Analysis Software (Becton Dickinson).

Group I:

Infliximab 5 mg/kg. i.v. at week 0, 2, 6, 14 and 22.

Group II:

Infliximab Placebo i.v. weeks 0, 2, 6, 14 and 22.

Extension Phase (weeks 24-48):

1. Responders at week 24: Treatment discontinuation (GROUP A).
2. No-responders at week 24:

   * Placebo group: infliximab (5 mg/kg) at weeks 24, 26, 30, 36 y 42 (GROUP B).
   * Infliximab group:
   * Patients who have lost response during phase 1 before week 24 will receive infliximab (5 mg/kg) at weeks 30, 36 and 42 (GROUP C).
   * Patients who never have fulfilled response criteria during Phase 1: will not receive treatment in extension phase. (GROUP D)

ELIGIBILITY:
Inclusion Criteria:

* PMR patients that after 2 years of corticosteroid treatment are not able to reduce the dose of prednisone below 5 mg/day or equivalent.
* PMR patients that after 6 months of corticosteroid treatment are not able to reduce the dose of prednisone below 7,5 mg/day or equivalent.
* PMR patients should fulfill the criteria proposed by Chuang et al (8):

  * Age ≥ of 50 years.
  * Development of bilateral moderately/severe aching and stiffness persisting for 1 month or more, involving two of the following areas: neck or torso, shoulders or proximal regions of the arms, and hips or proximal aspects of the thighs.
  * ESR ≥ 40 mm/h.
  * Complete clinical response to low-dose of steroids (prednisone or equivalent ≤ 20mg/day)

Exclusion Criteria:

* -Patients with biopsy-proven GCA or those with cranial symptoms or signs suggestive of GCA but without biopsy-proven arteritis.
* Patients with clinical features suggestive of RA or other connective tissue disorders.
* Chronic infections such as HIV, hepatitis B or C, active mycobacterial or fungal infections, etc.
* Neoplasm or a history of malignancy in the preceding 5 years.
* Patients with multiple sclerosis or other demilinizating disorders.
* Patients with cytopenias: leukopenia (leukocytes ≤ 3.5x109/L.), thrombocytopenia (platelets ≤ 100x109/L.) and/or anemia (≤ 10 g./dl.)
* Patients with cardiac failure (functional class III / IV).
* Any other condition that contraindicates Infliximab therapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2007-06; Primary Completion 2010-09 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of responders(complete remission without corticosteroids) | at 24 weeks

SECONDARY OUTCOMES:
Proportion of responders | at 48 weeks
Time to response | 48 weeks
Number of relapses / recurrences | 48 weeks
Response duration | 48 weeks
Cumulative dose and side effects of steroids | at 24 and 48 weeks
Number of patients that should be re-treated with infliximab | 48 weeks
Side effects of Infliximab in this patient population | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Víctor M Martínez-Taboada,, Md, PhD, Study Director — Servicio de Reumatología, Hospital Universitario Marques de Valdecilla; Vicente Rodriguez-Valverde, MD, PhD, Principal Investigator — Servicio de Reumatología, Hospital Universitario Marques de Valdecilla
Locations (1):
- Reumatology division, Hospital Universitario Marques de Valdecilla, Santander, Cantabria, Spain